CLINICAL TRIAL: NCT03571503
Title: The Effectiveness of Doin (Conduction Exercise) of the Pelvic Joint for Herniated Lumbar Disc (HLD) With Radiating Leg Pain: A Prospective Observational Pilot Study
Brief Title: The Effectiveness of Doin (Conduction Exercise) of the Pelvic Joint for HLD With Radiating Leg Pain
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, KIMMINYOUNG, Clinical Researcher, Jaseng Medical Foundation
Other Study IDs: JS-CT-2018-02
Record Dates: First submitted 2018-06-01; First posted 2018-06-27 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Intervertebral Disc Displacement; Sciatica; Sciatic Radiculopathy
Keywords: Complementary Therapies; Exercise; Acupuncture
MeSH Terms: conditions — Intervertebral Disc Displacement; Sciatica; Motor Activity | interventions — Phytotherapy; Acupuncture Therapy; Electroacupuncture; Cupping Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrative Korean medicine treatment: Herniated lumbar disc (HLD) patients with radiating leg pain in the integrative Korean medicine treatment group will be administered integrative Korean medicine treatment consisting of 2 sessions/day of acupuncture, and herbal medicine, Chuna manual therapy, bee venom pharmacopuncture and pharmacopuncture, electroacupuncture, cupping, and other interventions, as needed.
  Interventions: Drug: Herbal medicine; Procedure: Chuna manual therapy; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Other: Other intervention(s)
- Doin with integrative Korean medicine: Herniated lumbar disc (HLD) patients with radiating leg pain in the Doin (conduction exercise) with integrative Korean medicine treatment group will be administered integrative Korean medicine treatment consisting of 2 sessions/day of acupuncture, and herbal medicine, Chuna manual therapy, bee venom pharmacopuncture and pharmacopuncture, electroacupuncture, cupping, and other interventions, as needed, plus Doin (conduction exercise) for 1 session of the 2 sessions/day of acupuncture.
  Interventions: Procedure: Doin (conduction exercise); Drug: Herbal medicine; Procedure: Chuna manual therapy; Procedure: Bee venom pharmacopuncture; Procedure: Pharmacopuncture; Procedure: Acupuncture; Procedure: Electroacupuncture; Procedure: Cupping; Other: Other intervention(s)

INTERVENTIONS:
Procedure: Doin (conduction exercise) — An acupuncture physician will administer acupuncture at 4-8 acupoints in the low back and gluteal area (mandatory points: BL54, and GB30 ipsilateral to the dysfunctional site; and selective points: BL23, BL24, BL25, BL26, BL31, BL32, Ah-shi points, local acupuncture points and/or trigger points. Doin (conduction exercise) will be performed as active and passive movement with the needles in situ to the aim of effective treatment of pain and functional disability by increasing the hip joint range of motion (flexion and extension) with physician guidance and isometric resistance exercise (flexion and extension) as needed. Doin (conduction exercise) sessions will be performed 1 session/day for the duration of hospitalized treatment while the patient presents radiating leg pain (NRS≥1).
  Other Names: Doin Exercise; Do-in Exercise; Conduction Exercise
  Groups: Doin with integrative Korean medicine
Drug: Herbal medicine — Herbal medicine will be mainly administered in water-based decoction (120ml) and dried powder (2g) form (the ingredients are mainly, but not restricted to: Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes japonica, Psoralea corylifolia, Saposhnikovia divaricata, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, Glycine max, Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Chuna manual therapy — Chuna is a Korean spinal manipulation that incorporates spinal manipulation techniques for joint mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement. Chuna manipulation will be administered at the physician's discretion.
  Other Names: Chuna manipulation; Chuna spinal manipulation
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture will be administered only after confirming a negative response to hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) filtered for allergens will be injected at 4-5 acupoints proximal to the dysfunctional site at the physician's discretion. Each acupuncture point will be injected to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
  Other Names: Bee venom acupuncture
Procedure: Pharmacopuncture — Pharmacopuncture consisting of select herbal ingredients will be administered at Ah-shi points and local acupuncture points using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Acupuncture — Acupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Electroacupuncture — Electroacupuncture treatment will be administered using mainly proximal acupuncture points and Ah-shi points.
Procedure: Cupping — Cupping treatment will be administered at 1-2 points using mainly proximal acupuncture points and Ah-shi points.
Other: Other intervention(s) — Patients will be allowed any other additional intervention(s) as deemed necessary by the attending physician regardless of type or dose, and patterns of use will be investigated and recorded as an pragmatic clinical study.

SUMMARY:
A prospective pilot study will be conducted to investigate the effectiveness and safety in herniated lumbar disc (HLD) patients receiving integrative Korean medicine treatment including Doin (conduction exercise) at a Korean medicine hospital through assessment of pain, functional disability, and quality of life.

DETAILED DESCRIPTION:
A prospective single-center observational pilot study will be conducted to investigate the effectiveness and safety in herniated lumbar disc (HLD) patients with radiating leg pain receiving integrative Korean medicine treatment including Doin (conduction exercise) of the pelvic joint at Daejeon Jaseng Hospital of Korean Medicine through assessment of pain, functional disability, quality of life, satisfaction, and safety.

The study is expected to be performed over a period of 6 months, during the former 3 months of the study period of which the Integrative Korean medicine treatment group will be recruited, and after a wash-out period of 2 weeks, during the latter 3 months of the study period of which the Doin with integrative Korean medicine will be recruited separately.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with radiating leg pain distal to the gluteal fold with or without low back pain (LBP)
* Patients with onset of radiating leg pain occurrence within the last six months, and current pain intensity of numeric rating scale (NRS) ≥5
* Patients with disc protrusion or extrusion at the neural segment level with significant correlations with the radiating leg pain symptoms as identified on L-spine magnetic resonance imaging (MRI)
* Patients with plans of receiving Korean medicine treatment for herniated lumbar disc (HLD) through hospitalized care
* Patients who give voluntary written informed consent to study participation

Exclusion Criteria:

* Patients with other systemic diseases that may interfere with treatment effect or outcome interpretation
* Surgery and surgical procedure in the last three weeks in areas of clinical relevance as a result of HLD
* Patients with soft tissue pathologies or pathologies of non-spinal origin that may cause LBP or radiating leg pain (e.g. spinal tumor, rheumatoid arthritis)
* Patients for whom acupuncture treatment may be inappropriate or unsafe (e.g. hemorrhagic diseases, blood clotting disorders, history of anti-coagulation medicine intake, serious diabetes with risk of infection, severe cardiovascular diseases, or other conditions deemed unsuitable for acupuncture treatment)
* Pregnant patients or patients planning pregnancy
* Patients with serious psychological disorders
* Participating in other clinical studies other than observational studies
* Patients unable to fill out study participation consent form
* Subjects deemed unsuitable for study participation as assessed by the researchers

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Herniated lumbar disc (HLD) patients with radiating leg pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) of low back pain | Baseline, 2 weeks post-baseline
  Change in low back pain intensity at 2 weeks as measured using NRS. In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Change in Numeric Rating Scale (NRS) of radiating leg pain | Baseline, 2 weeks post-baseline
  Change in radiating leg pain intensity at 2 weeks as measured using NRS. In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Change in Oswestry Disability Index (ODI) | Baseline, 2 weeks post-baseline
  Functional disability questionnaire at 2 weeks as measured using ODI. The ODI is a 10-item questionnaire developed to assess level of disability due to low back pain (LBP). Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to LBP.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) of low back pain | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Low back pain intensity as measured using NRS. In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Numeric Rating Scale (NRS) of radiating leg pain | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Radiating leg pain intensity as measured using NRS. In pain measurement using NRS, patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Oswestry Disability Index (ODI) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Functional disability questionnaire as measured using ODI. The ODI is a 10-item questionnaire developed to assess level of disability due to low back pain (LBP). Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to LBP.
Visual Analogue Scale (VAS) of radiating leg pain | Baseline, 3, 7, 10, 14 days post-baseline
  Radiating leg pain intensity as measured using VAS. VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.
Visual Analogue Scale (VAS) of low back pain | Baseline, 3, 7, 10, 14 days post-baseline
  Low back pain intensity as measured using VAS. VAS uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain' and 'worst pain possible' (labels may vary by study). Scores are recorded in millimeters with a total range of 0-100 millimeters.
EuroQol 5-Dimension (EQ-5D) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Health-related quality of life questionnaire as measured using SF-36. SF-36 consists of 36 items across 8 domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. SF-36 is used to rate functional health and well-being in patients and healthy individuals. Higher scores indicate better HRQoL.
Patient Global Impression of Change (PGIC) | Baseline, 14, 30, 90 days post-baseline
  Global patient-reported outcome as measured using PGIC. PGIC grades the level of subjective improvement into 7 levels (1, very much improved; 2, much improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; and 7, very much worse).
Drug Consumption (drug type) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding recent use of medication, the type of prescription intake for medicine will be recorded.
Drug Consumption (drug intake frequency) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding recent use of medication, the frequency of prescription intake for medicine will be recorded.
Drug Consumption (drug intake period) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding recent use of medication, the period of prescription intake for medicine will be recorded.
Use of additional medical treatment (treatment type) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding current use of medical services, the type of additional medical treatment received will be recorded.
Use of additional medical treatment (treatment frequency) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding current use of medical services, the frequency of additional medical treatment received will be recorded.
Use of additional medical treatment (treatment period) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Regarding current use of medical services, the period of additional medical treatment received will be recorded.
Details of Doin conduction exercise sessions (type (region)) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Administration details of Doin conduction exercise session type (region) will be recorded.
Details of Doin conduction exercise sessions (period) | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Administration details of Doin conduction exercise sessions (period) will be recorded.
Lumbar range of movement (ROM) | Baseline, 3, 7, 10, 14 days post-baseline
  Physical examination
Straight leg raise (SLR) test | Baseline, 3, 7, 10, 14 days post-baseline
  Physical examination
Adverse events | Baseline, 3, 7, 10, 14, 30, 90 days post-baseline
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Min-young Kim, KMD, Principal Investigator — Daejeon Jaseng Hospital of Korean Medicine
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No